CLINICAL TRIAL: NCT03943368
Title: Using Virtual Reality (VR) Models for Robotic Prostatectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ceevra, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20171006RP
Record Dates: First submitted 2019-05-07; First posted 2019-05-09 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-06

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Experimental: Intervention Arm (Experimental): Subjects whose surgeon will be viewing Digital 3D models in addition to the source MR image and biopsy results in connection with the case.
  Interventions: Device: Ceevra Reveal
- Control Arm (No Intervention): Subjects whose surgeon will only be viewing MR images in connection with the case.

INTERVENTIONS:
Device: Ceevra Reveal — 3D Digital models generated using Ceevra Reveal are viewed by surgeons in connection with the case in addition to source MR image.
  Arms: Experimental: Intervention Arm

SUMMARY:
A prospective, randomized, controlled study designed to assess whether digital virtual reality (VR) models, created from existing CT scans and MRIs, provide surgeons with an improved understanding of their patients' anatomy, resulting in more efficient operations (robotic prostatectomy) and improved patient care.

ELIGIBILITY:
Inclusion Criteria:

* Patient is undergoing robotic prostatectomy being performed by participating surgeon
* Patient is willing to be randomized between intervention and control arms

Exclusion Criteria:

* Patients with prior pelvic radiation
* Patients with prior androgen deprivation therapy
* Patients with prior localized ablative therapy
* Patients with prior TURP or other surgical BPH treatment

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Postoperative PSA | Up to 24 months
  PSA blood test measured at threshold of 0.1 at 3-6 and 18-24 months

SECONDARY OUTCOMES:
Surgical Margin Status | Immediately postoperatively
  Defined as positive or negative surgical margin
Androgen Deprivation or Radiation Therapy | Up to 24 months postoperatively
  Any occurrence of salvage or adjuvant therapy post surgery
Postoperative Erectile Function | Up to 24 months postoperatively
  Nerve sparing immediately postoperatively, SHIM score at 3-6 and 18-24 months
Postoperative Urinary Function | Up to 24 months postoperatively
  Bladder neck sparing immediately postoperatively, pads per day at 3-6 and 18-24 months

CONTACTS AND LOCATIONS:
Overall Officials: James Porter, MD, Principal Investigator — Swedish Medical Center; Raymond Pak, MD, Principal Investigator — Mayo Clinic; Thomas Ahlering, MD, Principal Investigator — UC Irvine; Robert Reiter, MD, Principal Investigator — UCLA Urology; Ketan Badani, MD, Principal Investigator — Mount Sinai Health System
Locations (6):
- United States (6):
  - UCLA Urology, Los Angeles, California
  - UC Irvine, Orange, California
  - Mayo Clinic Florida, Jacksonville, Florida
  - Mount Sinai Health System, New York, New York
  - Swedish Urology Group, Seattle, Washington
  - Swedish Medical Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shirk JD, Reiter RE, Wallen EM, Pak RW, Ahlering T, Badani KK, Porter JR. Trifecta Outcomes After Use of 3-Dimensional Digital Models for Planning of Robotic Prostatectomy: A Secondary Analysis of a Randomized Clinical Trial. JAMA Netw Open. 2024 Sep 3;7(9):e2434143. doi: 10.1001/jamanetworkopen.2024.34143. PMID 39283633
- [Derived] Shirk JD, Reiter R, Wallen EM, Pak R, Ahlering T, Badani KK, Porter JR. Effect of 3-Dimensional, Virtual Reality Models for Surgical Planning of Robotic Prostatectomy on Trifecta Outcomes: A Randomized Clinical Trial. J Urol. 2022 Sep;208(3):618-625. doi: 10.1097/JU.0000000000002719. Epub 2022 Jul 18. PMID 35848770